CLINICAL TRIAL: NCT01927458
Title: Transcranial Direct Current Stimulation Aided Rehabilitation of Gait in Subacute Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Krystian Figlewski, MD, University of Aarhus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M-2012-570-12
Record Dates: First submitted 2013-08-15; First posted 2013-08-22 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Stroke; Neurorehabilitation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- anodal tDCS with treadmill training (Experimental): Each subject will receive 4 weeks gait treadmill training at least 3 days per week in combination with anodal transcranial Direct Current Stimulation over the primary motor cortex up to 20 min
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — A direct current runs between two electrode positions and affects the excitability of the underlying brain tissue
  Other Names: Non.invasive brain stimulation

SUMMARY:
The purpose of this study is to determine if transcranial direct current stimulation (tDCS)applied over the lower extremity motor cortex in conjunction with treadmill training is effective for improving gait in patients with subacute stroke and to evaluate the effect and predictive value of a single session of anodal tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Onset of stroke less than 14 days
* First ischemic stroke causing lower limb weakness (MRC score ≤4 in knee extensors) and gait impairment

Exclusion Criteria:

* Contraindications to MRI or TMS
* Other neurological disorders
* Significant somatic or psychiatric disorders
* History of seizures
* Language or cognitive disorders prohibiting participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximal gait speed using the 10-m walking test | Baseline and follow up immediately following the 4 weeks intervention

SECONDARY OUTCOMES:
Changes in cortical excitability measures | Baseline
  We will measure cortical excitability using single pulse transcranial magnetic stimulation (TMS) before and after 1st stimulation session. We will compare the measurements from before stimulation to after stimulation.
Dynamometry: the maximal isometric force of muscles will be assessed by Biodex System 3 PRO dynamometer | Baseline and immediately following the 4 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, Professor, Study Director — University of Aarhus
Locations (1):
- Hammel Neurocenter, Hammel, Denmark